CLINICAL TRIAL: NCT03384914
Title: A Multicenter Phase II Study of Vaccines to Prevent Recurrence in Patients With HER-2 Positive Breast Cancer
Brief Title: Vaccine to Prevent Recurrence in Patients With HER-2 Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19117
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Female; Breast Cancer, Male; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Residual Disease; HER2-positive Breast Cancer; HER2 Positive Breast Carcinoma
Keywords: axillary nodes; HER-2 directed treatment
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Neoplasm, Residual | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dendritic Cell (DC1) Vaccine (Active Comparator): The vaccine will be administered in two phases: a vaccination phase and a booster phase.
  Approximately 6 months from the initiation of the first vaccine, patients will receive the first of 3 booster vaccines.
  Interventions: Biological: DC1 Vaccine
- pUMVC3-IGFBP2-HER2-IGF1R (WOKVAC) (Active Comparator): The vaccine will be administered in two phases: a vaccination phase and a booster phase.
  Approximately 6 months from the initiation of the first vaccine, patients will receive the first of 3 booster vaccines.
  Interventions: Biological: WOKVAC Vaccine

INTERVENTIONS:
Biological: DC1 Vaccine — Vaccination Phase: DC1 vaccine will be administered weekly via intranodal injection in weeks 1 to 6 (window 8-21days between vaccines).
  Booster vaccines will be administered at approximately 3 month intervals on months 6, 9 and 12 (with a window +/- 1 month).
  Other Names: Immunotherapy; Dendritic Cell Vaccine
  Arms: Dendritic Cell (DC1) Vaccine
Biological: WOKVAC Vaccine — Vaccination Phase: WOKVAC vaccine will be administered via intradermal injection on weeks 1, 4 and 7 (window +21 days).
  Booster vaccines will be administered at approximately 3 month intervals on months 6, 9 and 12 (with a window +/- 1 month).
  Other Names: Immunotherapy; pUMVC3-IGFBP2-HER2-IGF1R
  Arms: pUMVC3-IGFBP2-HER2-IGF1R (WOKVAC)

SUMMARY:
The main purpose of this study is to evaluate the safety of each study vaccine and to evaluate the effect on the time to disease recurrence (assessed by disease free survival).

Participants will be assigned to receive one of two study vaccines (DC1 study vaccine vs. WOKVAC). The study vaccine will be administered in two phases: a study vaccination phase and a booster phase.

DETAILED DESCRIPTION:
The total duration of the study will be 6 years (4 years of patient enrollment and 2 additional years of clinical follow-up). Assessment for disease recurrence and survival will be conducted every 6 months (with a phone call/secure email, medical records or follow up visit) from the end of treatment for a total of 2 years, until the completion of the trial or until documented disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage I-III HER2 positive breast cancer treated with neoadjuvant chemotherapy including HER-2 directed treatment for at least 12 weeks.
* Residual invasive carcinoma in the breast or axillary nodes in the final pathology from resected tumor following neoadjuvant chemotherapy.
* Completed last cycle of cytotoxic chemotherapy (excluding ado-trastuzumab emtansine [T-DM1]) or radiation > 30 days with resolution of all acute toxic effects of prior therapy to grade ≤ 2 (except alopecia)
* Currently on HER-2 targeted therapy (eg; trastuzumab +/- pertuzumab or T-DM1) per standard of care or has completed HER-2 targeted therapy less than 6 months ago
* Age ≥ 18 years.
* Eastern Cooperative Group (ECOG) performance status 0 or 1.
* Must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,000/ μL
  * Platelets ≥ 75,000/ μL
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), except patients with Gilbert's syndrome in whom total bilirubin must be <3.0 mg/dL
  * AST/ALT ≤ 3 x institutional upper limit of normal (ULN)
  * Creatinine ≤ 1.5 x institutional upper limit of normal (ULN)
  * Hemoglobin A1C <6.5%
* Left ventricular ejection fraction (LVEF) above institutional lower limit of normal (by echocardiogram or MUGA scan within 90 days of registration).
* Females of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and males must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. For both male and female participants, effective methods of contraception must be used throughout the study and for three months following the last dose.
* Ability to understand and willingness to sign a written informed consent document prior to initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congenital prolonged QT syndrome, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Uncontrolled autoimmune disease requiring active systemic treatment.
* Known hypersensitivity reaction to the Granulocyte-macrophage colony stimulating factor (GM-CSF) adjuvant; any known contraindication to GM-CSF.
* Pregnant or breast feeding.
* Known HIV-positive.
* Known current or a history of hepatitis B or C virus, including chronic and dormant states, unless disease has been treated and confirmed cleared.
* Major surgery within 4 weeks of initiation of study drug.
* Current extended use of immunosuppressive agents or systemic corticosteroids. Topical, ocular, intra-articular, intranasal, inhalational corticosteroids (with minimal systemic absorption) are allowed. A brief course of corticosteroids for prophylaxis (eg., for contrast dye allergy) or for treatment of non-autoimmune conditions (eg., delayed-type hypersensitivity reaction caused by a contact allergen) is permitted.
* Potential participant is currently on active treatment in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices, or investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | Up to 3 years
  The primary immunogenicity outcome for both arms of this trial will be the summation of spots (ELISPOT) for 6 distinct peptides and reported as total SFC/10^6 cells. A value >150 defines an immune response.

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | Up to 3 years
  Clinical activity is characterized by disease-free survival (DFS), defined as the time from start of treatment to documented recurrence (any breast event), death due to any cause or last patient contact that documents recurrence-free status (i.e., a clinic or scan date).

CONTACTS AND LOCATIONS:
Overall Officials: Hyo S. Han, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (7):
- United States (7):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory - Winship Cancer Institute, Atlanta, Georgia
  - Indiana University - Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Ohio State University - Arthur G James Cancer Hospital & Richard J Solove Research Institute, Columbus, Ohio
  - University of Washington, Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/